CLINICAL TRIAL: NCT03157063
Title: Pilot Data Collection for Activity, Adiposity, and Appetite in Adolescents
Acronym: AAAA
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16120865
Record Dates: First submitted 2017-05-01; First posted 2017-05-17 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity; Sedentary Lifestyle; Metabolism; Energy Balance
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — hormones related to satiety and hunger (insulin, leptin, ghrelin, peptide YY, glucagon-like peptide-1) obtained during blood samples (BLOOD) from an indwelling catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Inactive, normal weight: Less than 30 minutes per day of moderate to vigorous physical activity (MVPA), and body mass index percentile (BMI%) between 5th to 75th percentile.
  Interventions: Diagnostic Test: Data Collection Procedures
- Inactive, overweight/obese: Less than 30 minutes per day MVPA, BMI% between 85th and 99th.
  Interventions: Diagnostic Test: Data Collection Procedures
- Active, normal weight: More than 60 minutes per day MVPA, BMI% between 5th and 75th.
  Interventions: Diagnostic Test: Data Collection Procedures
- Active, overweight/obese: More than 60 minutes per day MVPA, BMI% between 85th and 99th.
  Interventions: Diagnostic Test: Data Collection Procedures

INTERVENTIONS:
Diagnostic Test: Data Collection Procedures — Orientation (Consent, Screening Questionnaires) Clinic Measurements Body composition, via dual energy X-ray absorptiometry (DXA) Resting metabolic rate (RMR), via indirect calorimetry; Metabolic responses to a meal, via thermic effect of feeding (TEF) Subjective aspects of eating behavior using the Three Factor Eating Questionnaire (TFEQ) and Control of Eating Questionnaire (CEQ) Appetite, via visual analogue scales (VAS) pre- and post a prepared fixed meal and hormones related to satiety and hunger (insulin, leptin, ghrelin, peptide YY, glucagon-like peptide-1) obtained during blood samples (BLOOD) from an indwelling catheter.
  Home assessments - Data collected at home during a 14 day window Fitness Test (VO2submax and VO2max) and DXA functional magnetic resonance imaging (fMRI)

SUMMARY:
The goal of this study is to quantify energy metabolism using indirect calorimetry at rest, in the presence of excess energy following a meal, and in response to the demand for energy during exercise. The investigators also will examine the individual and joint associations of activity and obesity status on neurocognitive domains of appetite control. Participants will include adolescent males and females (N=80) using a 2 x 2 cross-sectional study design, stratified by body weight (normal vs overweight/obese) and physical activity level (sedentary vs. active).

DETAILED DESCRIPTION:
The investigators hypothesize that low levels of fitness and MVPA result in impaired metabolic function in adolescents. For this pilot study, the investigators will quantify variations in metabolic characteristics using a 2 x 2 cross-sectional study design, stratified by body weight (normal vs overweight/obese) and physical activity (sedentary vs. active). The goal is to identify metabolic factors that influence the energy balance system to directly inform interventions designed to prevent or reduce the prevalence of pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* Males (Tanner Stage III-IV), ages 14-18
* Weight stable (5% weight change) over the previous three months as assessed by self-report.
* BMI greater than 5th and less than 99th percentile
* Physically healthy for exercise as assessed by self report Physical Activity Readiness Questionnaire (PAR-Q) for children.
* For fMRI testing, all participants must be right handed and must have normal or corrected to normal vision (as they will be viewing pictures in the fMRI procedure).

Exclusion Criteria:

* History of restrained eating, eating disorders, bariatric surgery, or other significant medical diagnosis that could impact metabolism.
* Participants taking thyroid medications, beta blockers, or other stimulants (medications are known to affect physical activity level and metabolism).
* Due to fMRI procedure requirements, children with a history of Attention Deficit Hyperactivity Disorder (ADHD) or other diagnosed psychiatric issues will be excluded.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will include 60 adolescent males (aged 14-18 years, Tanner stages III- IV), equally enrolled based on physical activity and body weight status.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
The independent effects of physical inactivity and obesity on metabolic responses (energy expenditure) at rest, after a meal, and during exercise using indirect calorimetry. | 1 year
  The investigators will measure energy expenditure at rest (also called resting metabolic rate), following a fixed-calorie meal (also called thermic effect of feeding), and during submaximal walking on a treadmill, all using an indirect calorimeter.

SECONDARY OUTCOMES:
Physical activity levels, as measured by subjective appetite ratings and hormones related to appetite, independent of obesity status. | 2 years
  The investigators will measure subjective appetite ratings related to hunger, fullness, etc. using visual analog scales and hormones related to appetite control following a fixed-calorie meal and buffet-style meal.

OTHER OUTCOMES:
The neurocognitive mechanisms of appetite control as assessed by functional MRI. | 2 years
  The investigators will measure neural activity in reward (limbic) and self-control (prefrontal) areas of the brain using functional MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Shook, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
aggregate results will be shared

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03157063/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03157063/SAP_000.pdf